CLINICAL TRIAL: NCT06384534
Title: Exercise Performance on Ambient Air vs. Commonly Prescribed Nasal Low Oxygen Therapy - a Non-inferiority Trial in Patients With Exercise Induced Desaturation Due to Pulmonary Vascular Disease (PVD)
Brief Title: Exercise Performance on Ambient Air vs. Low-Flow Oxygen Therapy in Pulmonary Vascular Disease (PVD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PVD_6MWD_SOT
Record Dates: First submitted 2024-04-17; First posted 2024-04-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Vascular Disorder; Chronic Thromboembolic Pulmonary Hypertension; Pulmonary Arterial Hypertension
Keywords: Pulmonary Hypertension; Supplemental Oxygen Therapy; Pulmonary Arterial Hypertension; Chronic Thromboembolic Pulmonary Hypertension; Pulmonary Vascular Disease; 6 Minute Walking Distance
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Each participant is its own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambient air (Experimental): Patient will perform tests at University Hospital Zurich
  Interventions: Other: 6-minute walk distance (6MWD) test on ambient air
- SOT via basal canula (Active Comparator): Supplemental Oxygen Therapy (SOT) at approximately 3l/min will be provided via nasal canula from a small oxygen concentrator while the patient performs tests at University Hospital Zurich.
  Interventions: Other: 6-minute walk distance test with supplemental oxygen

INTERVENTIONS:
Other: 6-minute walk distance (6MWD) test on ambient air — 6-minute walk distance (6MWD) test will be performed on ambient air according to clinical standards
  Arms: Ambient air
Other: 6-minute walk distance test with supplemental oxygen — 6-minute walk distance (6MWD) test will be performed according to clinical standards additionally with supplemental oxygen therapy (approximately 3l/min, nasal)
  Arms: SOT via basal canula

SUMMARY:
The investigators aim to study the effect of SOT in Swiss residents with pulmonary vascular diseases (PVD) defined as pulmonary arterial hypertension (PAH) or chronic thromboembolic pulmonary hypertension (CTEPH).

DETAILED DESCRIPTION:
Participants with PVD diagnosed with precapillary PH with right heart catheterization and classified to groups 1 and 4 (PAH or CTEPH) who live in Switzerland will have 6-minute walk distance (6MWD) test with and without SOT approximately 3l/min via nasal cannula according to a randomized cross-over design.

The trial aims to test that the 6MWD with SOT is non-inferior to a 6MWD in the same participant under ambient air.

The effect size was estimated with a difference of less or equal to 35m compared under SOT compared to ambient air.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years of age
* Written informed consent
* Patients with diagnosed pulmonary arterial hypertension (PAH), distal chronic thromboembolic pulmonary hypertension (CTEPH)
* Former desaturation under exercise defined as Spo2-decrease >3%
* Treated with a stable drug therapy (with no changes for at least 14 days prior to screening)

Exclusion Criteria:

* Severe hypoxemia needing supplemental oxygen therapy defined as partial pressure of O2 (PaO2) < 6.9 Kilopascal (kPa)
* Pregnancy
* Unability or contraindications to undergo the investigated intervention
* Unability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
6-minute walk distance (6MWD) with supplemental oxygen therapy (SOT) vs. ambient air | after 6 minutes
  Change in 6MWD in meter between SOT via nasal cannula vs. ambient air

SECONDARY OUTCOMES:
SpO2 at rest and peak 6MWD with SOT vs. ambient air | after 6 minutes
  Change of the arterial oxygen saturation by pulse oximeter (SpO2) at rest and at peak 6MWD with SOT approximately 3l /min vs. ambient air
Heart rate at rest and peak 6MWD with SOT vs. ambient air | after 6 minutes
  Change of heart rate (bpm) at rest and at peak 6MWD with SOT vs. ambient air
Borg dyspnea atrest and peak 6MWD with SOT vs. ambient air | 6 minutes
  Change of Borg dyspnea scale (CR10, 0-10 where 10 is the worst dyspnea) at rest and at peak 6MWD with SOT vs. ambient air
Borg leg fatigue scale at rest and peak 6MWD with SOT vs. ambient air | 6 minutes
  Change of Borg leg fatigue scale (CR10, 0-10 where 10 is the strongest led fatugue) at rest and at peak 6MWD with SOT vs. ambient air
Blood pressure at rest and peak 6MWD with SOT vs. ambient air | after 6 minutes
  Change of Blood pressure (mmHg) at rest and at peak 6MWD with SOT vs. ambient air

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof. Dr., Principal Investigator — University Hospital Zurich, Department of Pulmonology
Locations (1):
- University Hospital Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided upon request and based on a clear intention reviewed by an ethical review board